CLINICAL TRIAL: NCT05389878
Title: STroke RehabilitATion REgistrY for Predicting Functional Outcomes
Brief Title: Implementation of a Registry for Patients with Stroke
Acronym: STRATEGY
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Francesca Cecchi, Principal Investigator, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: STRATEGY
Record Dates: First submitted 2022-02-23; First posted 2022-05-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Registry; Outcome; Predictors
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Stroke group: Patients with stroke addressing intensive inpatient rehabilitation, including and treatment, delivered according to an Individual Rehabilitation Project (IRP), defined according AHA ASA Stroke rehabilitation Guidelines (2016. The IRP was defined by an interdisciplinary team, coordinated by a physiatrist and designed according to patients' and caregivers' needs. The team included internists, physiotherapists, occupational therapists, nurses, speech therapists, and psychologists. The assessment protocol aimed to provide a reliable and synthetic assessment of patients' clinical conditions and function at admission and discharge. Each patient received at least three hours of specific rehabilitation per day. All patients received clinical observation and management, nurse management, physiotherapy. Speech, neuropsychological, and occupational therapy treatment were prescribed by physiatrist.
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — All patients addressing intemsive inpatient post stroke rehabilitation undergo a shared evidence based Integrated Care pathway that is routinely adopted in all the participating Centres

SUMMARY:
Pathology registers are scientific research tools for the development of epidemiological and clinical studies and health planning, which allows access to useful elements for planning adequate health services. The Registry collects demographic, clinical and functional data of stroke patients and arises from the need to order and update this information for epidemiological and research purposes, for a better knowledge of this pathology from a rehabilitation point of view and to accelerate the development of new treatments.

DETAILED DESCRIPTION:
The Italian Society of Physical and Rehabilitation Medicine has published a minimal assessment protocol for stroke patients1 (PMIC2020) to share the evaluation of stroke rehabilitation needs and outcomes at any time of the rehabilitation pathway, as grounds for a National Stroke Rehabilitation Registry (SRR).

The STRATEGY multicentric study aims to verify the feasibility of implementing a PMIC2020-based SRR in a routine clinical setting, and develop data-driven prognosis prediction models.

Demographic, functional and clinical variables will be collected at the admission and the discharge of the patient; in addition, two telephone follow-ups (three months and six months from the event) will be carried out

The study will involve several rehabilitation centers of the Don Gnocchi Foundation, Italy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years of age) with ischemic or haemorrhagic stroke, first event or with relapse, time to onset of stroke less than 6 months, signature of informed consent by the patient or family member.

Exclusion Criteria:

* Patients from Severe Acquired Brain Injuries units and / or with diseases that threaten the patient's life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke consecutively admitted in the centers involved
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in modified Barthel Index | Admission, discharge (average 30 days from admission), follow-up (6 months after stroke)
  measure of ability in activity of daily living range 0 worst- 100 best

SECONDARY OUTCOMES:
Change in modified Rankin Score | Admission, discharge (average 30 days from admission), follow-up (6 months after stroke)
  measure of global disability range 0 best-5 worst
Change in Functional Ambulation Category | Admission, discharge (average 30 days from admission), follow-up (6 months after stroke)
  measure of functional ambulation range 0 worst- 6 best
Change in Trunk Control Test | Admission, discharge (average 30 days from admission)
  measure of trunk control range 0 worst- 100 best
Change in Short Physical Performance Battery | Admission, discharge (average 30 days from admission)
  measure of lower limbs physical performance range 0 worst-12 best
Change in Motricity Index | Admission, discharge (average 30 days from admission)
  Measure of motricity in upper and lower limb range 0 worst-100 best
Change in Modified Ashworth Scale | Admission, discharge (average 30 days from admission)
  Measure of upper and lower limb spasticity range range 0 best 100
Change of Mini Mental State Examination | Admission, discharge (average 30 days from admission)
  Cogntive level, range from 0 worst - 30 best

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Cecchi, MD, Principal Investigator — IRCCS Fondazione don Carlo Gnocchi
Locations (4):
- Italy (4):
  - IRCCS Fondazione Don Carlo Gnocchi, Florence
  - IRCCS Fondazione Don Carlo Gnocchi Santa Maria Rinascente, Milan
  - Fondazione Don Gnocchi, Centro Santa Maria ai Servi, Parma
  - Fondazione Don Carlo Gnocchi Centro "Spalenza", Rovato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cecchi F, Cassio A, Lavezzi S, Scarponi F, Gatta G, Montis A, Bernucci C, Franceschini M, Bargellesi S, Paolucci S, Taricco M. Redefining a minimal assessment protocol for stroke rehabilitation: the new "Protocollo di Minima per l'ICtus" (PMIC2020). Eur J Phys Rehabil Med. 2021 Oct;57(5):669-676. doi: 10.23736/S1973-9087.21.06638-7. Epub 2021 May 27. PMID 34042407
- [Background] Cecchi F, Diverio M, Arienti C, Corbella E, Marrazzo F, Speranza G, Del Zotto E, Poggianti G, Gigliotti F, Polcaro P, Zingoni M, Antonioli D, Avila L, Barilli M, Romano E, Landucci Pellegrini L, Gambini M, Verdesca S, Bertolucci F, Mosca I, Gemignani P, Paperini A, Castagnoli C, Hochleitner I, Luisi ML, Lucidi G, Hakiki B, Gabrielli MA, Fruzzetti M, Bruzzi A, Bacci Bonotti E, Pancani S, Galeri S, Macchi C, Aprile I. Development and implementation of a stroke rehabilitation integrated care pathway in an Italian no profit institution: an observational study. Eur J Phys Rehabil Med. 2020 Dec;56(6):713-724. doi: 10.23736/S1973-9087.20.06195-X. PMID 33494558
- [Derived] Campagnini S, Sodero A, Baccini M, Hakiki B, Grippo A, Macchi C, Mannini A, Cecchi F. Prediction of the functional outcome of intensive inpatient rehabilitation after stroke using machine learning methods. Sci Rep. 2025 May 8;15(1):16083. doi: 10.1038/s41598-025-00781-1. PMID 40341247